CLINICAL TRIAL: NCT07066683
Title: Pilot Study to Evaluate Fatigue and Fatigability Profiles and Their Impact on Walking and Balance in Patients With Charcot-Marie-Tooth Type 1A Disease Using a Global Approach in Comparison to Healthy Volunteers.
Acronym: FatMobCMT1A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9161; 2024-A01500-47 (Other: ANSM)
Record Dates: First submitted 2025-03-19; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Charcot-Marie-Tooth Type 1A
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcot Marie Tooth type 1A (Experimental): CLINICAL ASSESSMENT OF BODY FUNCTION (PROM AND PHYSICAL EXAMINATION):
  * Perceived fatigue
  * Mental functions
  * Sensory functions and pain
  * Neuromusculoskeletal and movement-related functions
  * Functions of the cardiovascular and respiratory systems
    o Exercise stress test
  * Fatigability (neuromuscular fatigue)
    * Lower limbs
    * Maximum voluntary strength
    * Study of the central and peripheral components of fatigue
  ACTIVITIES AND PARTICIPATION
  * Mobility
    * Clinical standard tests for balance and walking
    * Quantified motion analysis
  * Activity level
  * Quality of life
  Interventions: Other: CLINICAL ASSESSMENT OF BODY FUNCTION (PROM AND PHYSICAL EXAMINATION) and ACTIVITIES AND PARTICIPATION
- Healthy subjects matched for age, height and lean body mass. (Active Comparator): Identical to patient, except for Charcot-Marie-Tooth specific tests
  Interventions: Other: CLINICAL ASSESSMENT OF BODY FUNCTION (PROM AND PHYSICAL EXAMINATION) and ACTIVITIES AND PARTICIPATION

INTERVENTIONS:
Other: CLINICAL ASSESSMENT OF BODY FUNCTION (PROM AND PHYSICAL EXAMINATION) and ACTIVITIES AND PARTICIPATION — Tip: Ensure that this name matches the name used in the associated Arm Description.
  CLINICAL ASSESSMENT OF BODY FUNCTION (PROM AND PHYSICAL EXAMINATION):
  * Perceived fatigue
  * Mental functions
  * Sensory functions and pain
  * Neuromusculoskeletal and movement-related functions
  * Functions of the cardiovascular and respiratory systems
    o Exercise stress test
  * Fatigability (neuromuscular fatigue)
    * Lower limbs
    * Maximum voluntary strength and power
    * Study of the central and peripheral components of fatigue
  ACTIVITIES AND PARTICIPATION
  * Mobility
    * Clinical standard tests for balance and walking
    * Quantified motion analysis
  * Activity level Quality of life The same evaluation tests will be performed on patients and healthy volunteer controls

SUMMARY:
Charcot-Marie-Tooth disease type 1A is the most common form of inherited neuropathy that causes peripheral nerve damage in all four limbs. In addition to the well-known distal motor and sensory symptoms, fatigue is one of the most common symptoms reported by patients. However, there is very little scientific data on this topic. Fatigue is associated with changes in mobility and quality of life. This study investigates the magnitude and impact of fatigue on patients' sensory-motor function and mobility (standing and walking). Fatigue is a complex phenomenon. It is therefore essential to assess all the factors that may be at the origin of this symptom (perceived fatigue and fatigability) using innovative and robust assessment methods.

These methods are based on quantitative non-invasive neurophysiologic measures (electromyography and transcranial magnetic stimulation). The patients can quantify and identify more precisely the origin of fatigability (peripheral and central). This objective approach needs to be combined with the usual methods of measuring fatigue using valid and reliable patient-reported outcome measures. A quantitative measure of movement during walking must also be included to assess changes in fatigue during functional movement.

To quantify the proportion of fatigue associated with CMT1A, the investigators chose to compare data from patients with those of healthy subjects matched for age, height and lean body mass.

A better understanding of the role of fatigue in limiting walking and balance capacities in these patients will allow the investigators to refine the inpatient and outpatient management.

ELIGIBILITY:
Inclusion criteria for patients:

* Age ≥ 18 years and < 75 years
* Patient with mCMT1A confirmed by genetic analysis (based on data recorded in the patient file)
* Patient able to walk a minimum of 200 metres without a break, with or without equipment and/or technical aids (collected during questioning)
* Patient able to get on and off a cycloergometer safely without assistance or with minimal assistance
* Patient who has had a cardiological check-up before the stress test (ECG and cardiac ultrasound less than 6 months old) or for whom a check-up is scheduled before the inclusion
* Patient affiliated to a health insurance scheme or beneficiary of such a scheme

Inclusion criteria for Healthy volunteers:

* Age ≥ 18 years and < 75 years
* Subject affiliated to or benefiting from a health insurance scheme
* Subject who has had a cardiological work-up prior to stress testing (ECG and cardiac ultrasound less than 6 months old) or for whom a work-up is scheduled prior to the procedure.

Exclusion criteria for patients:

* Patients with all other forms of neuropathy (HNPP, other types of CMT, secondary neuropathies)
* Patients with any of the following

  * An associated neurological disease other than mCMT1A
  * Severe joint disease of the lower limbs
  * Contraindication to isokinetic testing
  * Contraindication to an exercise stress test and exercise reconditioning program
  * A contraindication to Transcranial Magnetic Stimulation (TMS) : epilepsy, intracranial metallic foreign body, hearing aid or cochlear implant, unstable skull bone fracture, deafness, etc.
* Patients who have undergone lower limb surgery in the 12 months prior to inclusion or for whom lower limb surgery is scheduled during the participation period.
* Pregnant or breastfeeding or planning to become pregnant within the next 4 months
* BMI > 35 kg/m2
* Patient unable to give informed consent, unable to understand informed information
* Subject under court protection
* Subject under guardianship or curatorship
* Subject in a period of exclusion (determined by a previous or current study)

Exclusion criteria for healthy volunteers:

* History of neurological disease
* Severe joint damage in the lower limbs
* Any of the following

  * Contraindication to isokinetic testing
  * A contraindication to an exercise stress test and an exercise reconditioning program
  * A contraindication to TMS: epilepsy, intracranial metallic foreign body, hearing aid or cochlear implant, unstable skull bone fracture, deafness, etc.
* Any person who has undergone surgery on the lower limbs in the 12 months prior to inclusion, or for whom surgery on the lower limbs is scheduled during the participation period.
* Pregnant or breastfeeding, or planning to become pregnant within the next 4 months
* Person unable to give informed consent, unable to understand informed information
* BMI > 35 kg/m2
* Person under legal protection
* Person under guardianship or curatorship
* Person in a period of exclusion (determined by a previous or current study)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fatigability profile | 7 days
  Difference in isometric force developed by the knee extensors (assessment of overall neuromuscular fatigue) before and after a tiring exercise (stress test), during a maximum voluntary contraction, expressed in N.m-1, assessed on an isokinetic dynamometer (CONTREX®), compared between patients with mCMT1A and healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle de médecine physique et de réadaptation, Hôpital de Hautepierre, Strasbourg Centre de référence des maladies neuromusculaires, Institut Universitaire de Réadaptation Clémenceau, Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided